CLINICAL TRIAL: NCT00161655
Title: A Multicenter, Open-label, Randomized, Pilot-study to Evaluate the Efficacy and Safety of the Combination of Etanercept (ETN) and Methotrexate and of Etanercept (ETN) Alone in Patients With Plaque Psoriasis Despite Methotrexate Therapy
Brief Title: Study Evaluating Etanercept and Methotrexate in Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A-101696
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Psoriasis; Arthritis, Psoriatic
Keywords: Psoriasis; Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Arthritis | interventions — Etanercept; Methotrexate

INTERVENTIONS:
Drug: Etanercept
Drug: Methotrexate

SUMMARY:
The purpose of this study is to evaluate the efficacy to clear or almost clear the plaques in plaque psoriasis patients, treated with the combination etanercept and methotrexate compared to etanercept alone.

ELIGIBILITY:
Inclusion Criteria:

* Active plaque psoriasis involving >10% body surface area and/or minimal screening PASI score 8.
* Methotrexate >7.5 mg/week for the last 3 months

Exclusion Criteria:

* Predominantly guttate, erythrodermic or pustular psoriasis
* Other skin conditions than psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Primary Completion 2006-08 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Proportion of pts whose plaque psoriasis is cleared or almost cleared after 24 weeks.

SECONDARY OUTCOMES:
Percentage improvement in PASI. Proportion of pts demonstrating PASI 50, 75
and 90. Time to clear or almost clear on PGA.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (8):
- Denmark (2):
  - Fredriksberg Alle, Copenhagen
  - Gentofte Amtsygehus, Hellerup
- Finland (2):
  - Helsinki, Helsinki
  - Tampere, Pirkanmaa
- Norway (2):
  - Rikshospitalet, Olso
  - Hudlegekontoret Akutten, Tromso
- Sweden (2):
  - Lakarhuset Fasta Centrum, Farsta
  - Lakarhuset, Vallingby